CLINICAL TRIAL: NCT00001827
Title: Vaccine Therapy With Tumor Specific p53 Peptides in Adult Patients With Low Burden Adenocarcinoma of the Ovary
Brief Title: p53 Vaccine for Ovarian Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 990137; 99-C-0137; NCT00019903 (obsolete NCT alias)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2013-01-25

CONDITIONS: Ovarian Neoplasm
Keywords: Immunotherapy; Cancer; Oncogenes; T-cells; Vaccine Therapy; p53 Peptide; Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms | interventions — aldesleukin; incomplete Freund's adjuvant; p53 synthetic long peptide vaccine; sargramostim

INTERVENTIONS:
Biological: aldesleukin
Biological: incomplete Freund's adjuvant
Biological: p53 peptide vaccine
Biological: sargramostim
Biological: therapeutic autologous dendritic cells
Procedure: in vitro-treated peripheral blood stem cell transplantation

SUMMARY:
This study will examine whether vaccination with a p53 peptide can boost an immune response to ovarian cancer and what the side effects are of the vaccine.

Many patients with ovarian cancer have an altered (mutated) gene called p53 that causes the production of abnormal proteins found in their tumor cells. The body s immune system may try, unsuccessfully, to fight these abnormal proteins. In this study, ovarian cancer patients with a p53 abnormality will be vaccinated with a p53 peptide a part of the same abnormal protein found in their tumor to try to boost their body s immune response to the cancer.

Patients will be divided into two groups. Group A will have four p53 peptide vaccinations three weeks apart, injected under the skin. The injection will include a drug called ISA-51, which increases the effect of the vaccine. This group will also receive two other drugs that boost the immune system, IL-2 and GM-CSF. Group B will have four p53 peptide vaccinations three weeks apart. The peptide will be mixed with the patient s own blood cells and infused into a vein. This group will also receive IL-2, but not GM-CSF.

All study candidates will be tested to see if their cancer has a p53 abnormality and if their immune system mounted a defense against it. These tests may include a tumor biopsy (removal of a small part of the tumor for microscopic examination); lymphapheresis (a procedure to take blood, remove white blood cells called lymphocytes, and return the red cells); and an immune response test similar to a skin test for tuberculosis. During the study, patients will have additional skin tests and blood tests.

DETAILED DESCRIPTION:
P53 is the most commonly mutated gene in human cancers; it has been found to be mutated in almost 50% of ovarian cancers. Genetic mutation of p53 results in stabilization and increase in the level of the protein. In some cases, overexpression of p53 protein could also occur in tumors without detectable mutation in the open reading frame. Therefore, p53 could function as an antigen through two different mechanisms, as a mutant "foreign" protein and as a selfoverexpressed protein. The p53:264 - 272 wild type peptide has been shown to have high affinity for HLA-A2. It has also been shown to be naturally processed and endogenously

presented by HLA-A2 in different types of tumor cell lines for CTL recognition. These CTL

were able to lyse tumor cells overexpressing wild type or mutant p53 protein and failed to lyse

normal cells expressing normal levels of wild type p53.

In this protocol we will be vaccinating HLA-A2+ ovarian cancer patients who carry tumors which overexpress p53 with the wild type p53 peptide (264-272). This will be given either subcutaneously admixed with ISA-51 and GM-CSF adjuvants, or intravenously pulsed on dendritic cells along with low dose subcutaneous IL-2. In addition, those patients who express mutant p53 may also be vaccinated with a mutant p53 peptide, which corresponds to the mutation they harbor in their tumor, should the patients progress on the p53 (264-272) peptide.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must be 18 years of age or older.

Histologic diagnosis of adenocarcinoma of the ovary.

Tumor tissue availability for determination of p53 protein expression and genetic mutation (paraffin block, or fresh tissue).

Immunohistochemical analysis of the tumor must demonstrate positive p53 staining.

Patients should have ovarian cancer with marker only disease or patients with stage III, IV or recurrent who are NED post therapy.

ECOG performance status of 1 or 0.

Expected survival of more than 3 months.

The patients should not have received chemotherapy, radiation therapy, immunotherapy or systemic doses of steroids for at least 4 weeks prior to starting vaccination. And the patient should have recovered from all acute toxicities of previous treatment. Patients who received bone marrow transplantation within a year will not be eligible for the trial.

Patients must understand and sign an informed consent document that explains the neoplastic nature of his/her disease, the procedures to be followed, the experimental nature of the treatment, alternative treatments, and potential risks and toxicities.

Patients should have HLA-A2.1 haplotype.

EXCLUSION CRITERIA:

Any condition that does not fit with the eligibility criteria.

Any of the following:

Platelets less than 100K/mm(3)

Creatinine greater than 2.0 mg/dl

Serum Bilirubin greater than 2.0 mg/dl, SGOT, or SGPT greater than 4 times normal

HIV or Hepatitis B or C (i.e. detectable HBS Antigen or HC Ab) since these conditions might have an effect on the immune system.

Pregnant women or nursing mothers are ineligible since the effect of this investigational treatment on the health of the embryo is not known. Women with reproductive potential must have negative pregnancy test and must use adequate contraception.

Patients with active ischemic heart disease (i.e. Class III or IV cardiac disease-New York Heart Association), a recent history of myocardial infarction (within the last 6 months), history of congestive heart failure, ventricular arrythmias or other arrythmias requiring therapy.

Second malignancy (within the past 2 years) other than curatively treated carcinoma in-situ of cervix or basal cell carcinoma of the skin. These patients will be excluded for the possibility of the existence of a different mutation in the other primary malignancy.

History of CNS metastases.

Patients with underlying immune deficiency or history of autoimmune disease e.g. (autoimmune neutropenia, thrombocytopenia, or hemolytic anemia; systemic lupus erythematosus, Sjogren syndrome, or scleroderma; myasthenia gravis; Goodpasture syndrome; Addison's disease, Hashimoto's thyroiditis, active Graves' disease, or other diseases which qualify as autoimmune in origin).

Patients with active infections requiring antibiotics. Patients requiring chronic suppressive antibiotics will be eligible for the trial.

If, in the opinion of the principal or associate investigators, it is not in the best medical interest of the patient to enter this study, the patient will be ineligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 1999-07-26; Primary Completion 2007-12-17 (Actual); Study Completion 2013-01-25 (Actual)

PRIMARY OUTCOMES:
Cellular immunity as measured by Elispot assay and 51 Cr-release assay at baseline and every 3 weeks.

SECONDARY OUTCOMES:
Toxicity as measured by Common Toxicity Criteria v2.0 at baseline and every 3 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jay A Berzofsky, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Takahashi H, Merli S, Putney SD, Houghten R, Moss B, Germain RN, Berzofsky JA. A single amino acid interchange yields reciprocal CTL specificities for HIV-1 gp160. Science. 1989 Oct 6;246(4926):118-21. doi: 10.1126/science.2789433.
- [Background] Chiba I, Takahashi T, Nau MM, D'Amico D, Curiel DT, Mitsudomi T, Buchhagen DL, Carbone D, Piantadosi S, Koga H, et al. Mutations in the p53 gene are frequent in primary, resected non-small cell lung cancer. Lung Cancer Study Group. Oncogene. 1990 Oct;5(10):1603-10. PMID 1979160
- [Background] Mitsudomi T, Steinberg SM, Nau MM, Carbone D, D'Amico D, Bodner S, Oie HK, Linnoila RI, Mulshine JL, Minna JD, et al. p53 gene mutations in non-small-cell lung cancer cell lines and their correlation with the presence of ras mutations and clinical features. Oncogene. 1992 Jan;7(1):171-80. PMID 1311061